CLINICAL TRIAL: NCT00261261
Title: Study of the ADVANCE Behavioral Preparation Program for Children and Their Parents
Brief Title: Family-Centered Behavioral Preparation for Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ADVANCE
Record Dates: First submitted 2005-11-30; First posted 2005-12-02 (Estimated); Last update posted 2005-12-02 (Estimated); Status verified 2005-11

CONDITIONS: Anxiety
Keywords: children; anxiety; behavioral preparation; family; surgery; parents
MeSH Terms: conditions — Anxiety Disorders | interventions — Midazolam

INTERVENTIONS:
Behavioral: ADVANCE
Drug: Midazolam
Procedure: Parental presence

SUMMARY:
Children experience significant anxiety and distress during the preoperative period. Currently available interventions are ineffective and/or associated with significant disadvantages. These interventions exclusively target the child and do not attempt to reduce parental anxiety. Based on an integration of the literature in both the anesthesia and psychological milieus, we developed ADVANCE, a behaviorally oriented anxiety reduction program for children undergoing surgery that targets the family as a whole.

DETAILED DESCRIPTION:
Children and their parents (n=408) were randomly assigned to one of four groups: 1) Control: received standard of care, 2) PPIA: received standard parental presence during induction of anesthesia, 3) ADVANCE: received family-centered behavioral preparation, and 4) oral Midazolam. We assessed the effect of group assignment on anxiety levels and postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Children 2-10 years old who were in good health (American Society of Anesthesiology physical status I-II) and who were undergoing general anesthesia and elective, outpatient surgery, and their parents.

Exclusion Criteria:

* Children with a history of chronic illness, prematurity (fewer than 36 weeks gestation) or reported developmental delay

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400
Dates: Start 2001-01; Study Completion 2004-12

PRIMARY OUTCOMES:
Anxiety in children: modified Yale Preoperative anxiety scale
Anxiety in parents: STAI

SECONDARY OUTCOMES:
Emergence delirium
Analgesic consumption
Time to discharge from recovery room

CONTACTS AND LOCATIONS:
Overall Officials: Zeev N Kain, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States